CLINICAL TRIAL: NCT03680495
Title: Targeting Steroid Resistance During Acute Exacerbations of Chronic Obstructive Pulmonary Disease With Respiratory Failure - The AECOPD Resistance Study
Brief Title: Steroid Resistance During COPD Exacerbations With Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0256
Record Dates: First submitted 2018-06-21; First posted 2018-09-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: COPD; Emphysema or COPD; COPD Exacerbation; COPD Exacerbation Acute; Respiratory Failure; Ventilatory Failure
Keywords: COPD; Steroid Resistance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Respiratory Insufficiency; Hypoventilation | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Collection of whole blood, serum, plasma, PBMCs, urine, nasal cells, and microbiome from the mouth, sinonasal passage, lung and stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- AECOPD with Respiratory Failure: The AECOPD cohort will be hospitalized for an acute exacerbation of chronic obstructive pulmonary disease (AECOPD) with respiratory failure requiring invasive or non-invasive mechanical ventilation. We will be following patients from admission through to discharge, and during a follow-up visit (~2 months from discharge). During the follow-up visit we will be administering 60mg of methylprednisolone once to study possible steroid resistance.
  Interventions: Drug: Methylprednisolone
- Stable COPD: The Stable COPD cohort will not have had an AECOPD within the past 6 months and will be frequency matched to the AECOPD cohort. The Stable COPD cohort will have one research visit where we will administer 60mg of methylprednisolone once to study possible steroid resistance.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — 1. Methylprednisolone is a steroid (corticosteroid) similar to a product produced in the adrenal glands. It is used to help relieve inflammation (swelling, heat, redness, and pain) and is used to treat certain medical issues including COPD.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a lung disease caused by cigarette smoke that affects millions of people. In the United States, COPD is the 3rd leading cause of death making it one of our most important public health problems. Some people with COPD get disease flares that are called acute exacerbations of COPD - or AECOPDs for short. When people get an AECOPD they experience increased shortness of breath, wheezing and cough; symptoms that often require urgent or emergent treatment by healthcare providers. In the most severe, life-threatening situations, people with AECOPDs are put on a ventilator in the emergency department and admitted to the intensive care unit. Most AECOPDs can be treated with low doses of medications called steroids. This is good because high doses of steroids can cause unwanted side effects. Unfortunately, recent studies suggest that the sickest people, those admitted to the intensive care unit needing ventilator support, need higher doses of steroids because they may have resistance to these important medications. The investigators are studying steroid resistance during very severe AECOPDs so that we can eventually develop better and safer therapies for these vulnerable people.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a cigarette smoke-induced disease of the lungs that affects millions of people in the United States and worldwide. COPD is the 3rd leading cause of death, making it one our most important public health problems. Perhaps most importantly, COPD confines many people to their homes, tethers them to oxygen lines, and destroys their independence. Like many diseases of chronic inflammation, the course of COPD is marred by intermittent disease flares that need more intensive treatment. In COPD, disease flares are called acute exacerbations of COPD (AECOPDs). AECOPDs are characterized by increased shortness of breath, wheezing or cough that leads to urgent, and sometimes emergent, treatment with inhaled bronchodilators, antibiotics and steroids. AECOPDs can be devastating to many because they worsen quality of life and lung function, frequently lead to hospitalization, and increase the risk of death. For instance, the death rate can reach 25-30% when COPD patients are admitted to the intensive care unit with respiratory failure (i.e. needing ventilator support). Accordingly, our research is focused on improving outcomes in the sickest patients admitted to the hospital with an AECOPD.

Oral or intravenous steroids (glucocorticoids) have been the mainstay of treatment for over 40 years, but virtually no research has been done to determine the optimal therapy for the sickest patients who are admitted to the intensive care unit. Results from the few clinical studies suggest that steroid resistance is increased in these critically-ill patients and that many physicians under- or over-dose steroids. For example, patients hospitalized with an AECOPD (without respiratory failure) are effectively treated with steroids (such as prednisone) dosed as low as 40mg/day. In contrast, two recent clinical studies showed that ~80mg/day of prednisone was ineffective for AECOPD patients hospitalized with respiratory failure (those who require ventilatory support), while in a second study ~160mg/day of methylprednisolone improved outcomes. The investigators recent epidemiologic study showed that 66% of patients admitted with an AECOPD and respiratory failure between 2003-2008 were treated with >240mg/day of methylprednisolone, a dose that increases steroid-related side effects. The investigators hypothesize that there is a stepwise increase in steroid resistance with COPD<AECOPD<AECOPD with respiratory failure. A newly launched team of investigators is focused on establishing the presence of steroid resistance, defining the cause(s), devising new treatments to combat this problem and optimizing therapy for these vulnerable patients.

Steroids suppress inflammation by inducing anti-inflammatory genes, such as the dual-specificity phosphatase (DUSP) family - including DUSP1. DUSP1 inhibits inflammatory cytokines by removing phosphates from p38 and c-Jun N-terminal kinase (JNK) mitogen-activated protein kinases, which turns them off. Preliminary data show that DUSP1 is decreased in alveolar macrophages from COPD patients, suggesting the central hypothesis that steroid resistance is increased in AECOPDs with respiratory failure due to impaired glucocorticoid-mediated induction of DUSP1. To address this hypothesis, the investigators will inject 23 AECOPD patients with respiratory failure and 23 matched stable COPD subjects with 60mg of methylprednisolone to: 1) determine the presence of corticosteroid resistance in AECOPDs, 2) determine the role of DUSP1, and 3) examine alternative mechanisms driving steroid resistance. The goal of The AECOPD Resistance Study is to identify targets associated with steroid resistance in AECOPDs with respiratory failure to pave the way for new treatments based upon novel mechanisms.

ELIGIBILITY:
Inclusion Criteria for AECOPD with Ventilatory Failure Cohort:

* Emergency Department (ED) or ICU physician diagnosis of an acute exacerbation of COPD
* Age ≥ 40 years of age
* Need for ventilator support in the ED or ICU during the first 24 hours

Inclusion Criteria for Stable COPD Cohort:

* Physician diagnosis of COPD
* Age ≥ 40 years of age
* Frequency matched to AECOPD subjects for:

  * Age (± 10 year increments)
  * Current/Former smoking status (former smoker = no smoking for ≥ 1 month)
  * Lung function (FEV1% predicted by ± 10% increments)

Exclusion Criteria for AECOPD with Ventilatory Failure Cohort:

* Systemic steroid use ≤ 30 days prior to return visit
* Infection requiring antibiotics ≤ 1 month prior to return visit
* Hemoglobin < 8.0 g/dl
* Acute pulmonary embolism
* Diabetes
* History of immunodeficiency, interstitial lung disease, neuromuscular disorder or heart failure with respiratory exacerbation
* Tracheostomy
* Drugs that induce cytochrome P450 3A enzyme activity (e.g. barbiturates, phenytoin or carbamazepine) or drugs that inhibit cytochrome P450 3A activity (e.g. ketoconazole and chronic macrolide antibiotics)
* Age ≥ 90 year of age
* Known pregnancy
* Nursing mothers
* Prisoners

Exclusion Criteria for Stable COPD Cohort:

* Systemic steroid use ≤ 30 days prior to return visit
* Infection requiring antibiotics ≤ 1 month prior to return visit
* Hemoglobin < 8.0 g/dl
* Acute pulmonary embolism
* Diabetes
* History of immunodeficiency, interstitial lung disease, neuromuscular disorder or heart failure with respiratory exacerbation
* Tracheostomy
* Drugs that induce cytochrome P450 3A enzyme activity (e.g. barbiturates, phenytoin or carbamazepine) or drugs that inhibit cytochrome P450 3A activity (e.g. ketoconazole and chronic macrolide antibiotics)
* Age ≥ 90 year of age
* Known pregnancy
* Nursing mothers
* Prisoners

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The AECOPD Cohort will be selected from University of Colorado Hospital inpatient units during an exacerbation of their COPD requiring respiratory failure.
  The COPD Cohort will be selected from the pulmonary clinics at the University of Colorado Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Presence of steroid resistance in patients recently admitted with an acute exacerbation of chronic obstructive pulmonary disease with respiratory failure. | Once at ≥ 45 days after hospital discharge
  The ability of methylprednisolone to suppress interleukin-8 (IL-8) release from lipopolysaccharide (LPS)-stimulated peripheral blood mononuclear cells (PBMCs).

SECONDARY OUTCOMES:
Expression of Dual Specificity Phosphatase 1 (DUSP1) | Once at ≥ 45 days after hospital discharge
  Baseline expression and induction of Dual Specificity Phosphatase 1 (DUSP1) in peripheral blood monocytes from patients recently admitted with an acute exacerbation of chronic obstructive pulmonary disease with respiratory failure versus stable, matched controls.
Activity of the Mitogen-activated Protein (MAP) Kinase Pathway. | Once at ≥ 45 days after hospital discharge
  Differences in Mitogen-activated Protein (MAP) Kinase Pathway activity in peripheral blood monocytes from patients recently admitted with an acute exacerbation of chronic obstructive pulmonary disease with respiratory failure versus stable, matched controls.
Expression of Glucocorticoid-induced leucine zipper (GILZ) and DUSP Isoforms. | Once at ≥ 45 days after hospital discharge
  Baseline expression and induction of Glucocorticoid-induced Leucine Zipper (GILZ) and DUSP isoforms in peripheral blood monocytes from patients recently admitted with an acute exacerbation of chronic obstructive pulmonary disease with respiratory failure versus stable, matched controls.
Role of Phosphoinositide 3-kinase (PI3K) and Histone Deacetylase 2 (HDAC2) in steroid resistance. | Once at ≥ 45 days after hospital discharge
  The role of HDAC2 in steroid resistance will be examined by measuring HDAC2 expression and histone transacetylase and deacetylase activity in PBMCs.
Methylprednisolone pharmacokinetics following an acute exacerbation of chronic obstructive pulmonary disease with respiratory failure. | Once at ≥ 45 days after hospital discharge
  Measuring methylprednisolone pharmacokinetics in patients following an acute exacerbation of COPD with respiratory failure versus a stable, matched control.
Examination of steroid-responsive gene expression patterns following an acute exacerbation of COPD with respiratory failure. | Once at ≥ 45 days after hospital discharge
  Ribonucleic acid (RNA) sequencing will be performed on PBMCs from patients and controls before and after exposure to methylprednisolone.

CONTACTS AND LOCATIONS:
Overall Officials: William Vandivier, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided